CLINICAL TRIAL: NCT03508154
Title: Evaluation of Carbohydrates: Glycemic Index of Nutrition Product Formulation
Brief Title: Evaluation of Carbohydrates - Glycemic Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DA19
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Meal 1 (Active Comparator): Control carbohydrate solution
  Interventions: Other: Control Meal 1
- Control Meal 2 (Active Comparator): Control carbohydrate solution
  Interventions: Other: Control Meal 2
- Experimental Nutritional Product (Experimental): Study nutritional formulation
  Interventions: Other: Experimental Nutritional Product

INTERVENTIONS:
Other: Control Meal 1 — carbohydrate test meal
  Arms: Control Meal 1
Other: Control Meal 2 — carbohydrate test meal
  Arms: Control Meal 2
Other: Experimental Nutritional Product — ready to drink nutritional formulation
  Arms: Experimental Nutritional Product

SUMMARY:
This study is an open-label with a randomized, cross-over design using standard GI methodology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are males or non-pregnant females in good health
* Subjects must be eligible to receive income in Canada and must demonstrate OHIP or equivalent medical coverage.

Exclusion Criteria:

* Subjects with any type of food allergy or known history of AIDS, hepatitis, diabetes or a heart condition
* Subjects taking medication, or with any condition which might, in the opinion of the PI either make participation dangerous to the subject or to others or affect the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Blood glucose response curve | 0 to 120 minutes
  area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dumas, Study Chair — Abbott Nutrition
Locations (1):
- Glycemic Index Laboratories Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided